CLINICAL TRIAL: NCT05019859
Title: Effects of a Low Carb Diet on Erectile Function and Serem Testosterone in Men With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMoinhosVento
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2021-07

CONDITIONS: Testosterone Deficiency; Metabolic Syndrome; Diet Modification
Keywords: low carb diet; hypogonadism; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Hypogonadism

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): low carb diet
  Interventions: Behavioral: low carb diet
- Control (No Intervention): traditional low fat diet

INTERVENTIONS:
Behavioral: low carb diet — low carb diet
  Arms: Intervention

SUMMARY:
Investigate if low carb diet could increase serum testosterone level in hypogonadic men

DETAILED DESCRIPTION:
Randomized controlled trial to evaluate the effect of low carb diet in men with metabolic syndrome and low testosterone level. The inclusion criteria is men with metabolic syndrome and serum total testosterone below 300 ng/dL. They will randomized to perform a low carb diet or a traditional low fat diet for metabolic syndrome. The follow up will be of three months with a once a month visit. Even though these men will be looked at their sexuality and life style. They will be monitoring by urologists and nutritionists during the study.

ELIGIBILITY:
Inclusion Criteria:

* metabolic syndrome, serum testosterone level below 300 ng/dL

Exclusion Criteria:

* active cancer, diet allergies, psychological incapability

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
testosterone | three months
  serum total testosterone level

SECONDARY OUTCOMES:
IIEF 5 | three months
  International Index of Erectile Function 5
AMS | three months
  Age male Symptom score

CONTACTS AND LOCATIONS:
Overall Officials: Brasil S Neto, MD, PhD, Study Chair — Hospital de Clínicas Porto Alegre; Caio S Schmitt, MD, Principal Investigator — Hospital Moinhos de Vento and Hospital de Clínicas Porto Alegre
Locations (1):
- Hospital de Clínicas Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil